CLINICAL TRIAL: NCT07353892
Title: Robotic Exoskeletons in Acute Care Therapy - Cardiovascular and Thoracic Surgery
Brief Title: Robotic Exoskeletons in Acute Care Therapy
Acronym: REACT-CVTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 025-408
Record Dates: First submitted 2025-12-04; First posted 2026-01-21 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Patients Post-cardiothoracic Surgery
Keywords: cardiothoracic surgery; rehabilitation; ambulation

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to experimental treatment vs. Standard -of care treatment in 2:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Overground robotic exoskeleton early ambulation (ORE-EA) (Experimental): Overground robotic exoskeleton early ambulation (ORE-EA)
  Interventions: Device: Overground robotic exoskeleton early ambulation (ORE-EA)
- Usual care early ambulation (UC-EA) (Active Comparator): Standard of care
  Interventions: Other: Usual care early ambulation (UC-EA)

INTERVENTIONS:
Device: Overground robotic exoskeleton early ambulation (ORE-EA) — Overground robotic exoskeleton early ambulation (ORE-EA)
  Arms: Overground robotic exoskeleton early ambulation (ORE-EA)
Other: Usual care early ambulation (UC-EA) — Usual care early ambulation (UC-EA) program for rehabilitation
  Arms: Usual care early ambulation (UC-EA)

SUMMARY:
The goal of this clinical trial is to establish the safety, feasibility, and preliminary findings of overground robotic exoskeleton early ambulation (ORE-EA) compared to usual care early ambulation (UC-EA) in the rehabilitation of patients who have had cardiovascular or thoracic surgery. The main questions it aims to answer are:

* Is there a difference between groups in time between surgery and ambulation?
* Are there differences in safety and feasibility?

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Underwent cardiovascular or thoracic surgery, including but not limited to coronary artery bypass grafting, valve replacement/repair, lung resection, or advanced cardiovascular or pulmonary therapies [transplant, durable or temporary ventricular assist device implantation (VAD), temporary mechanical circulatory support (tMCS), venovenous extracorporeal membrane oxygenation (VV ECMO)].
3. Medically appropriate for physical therapy, including upright activity and ambulation, as defined by an order in the patient's electronic medical record signed by a physician or advanced practice provider.
4. Requires ≥ 50% assist to perform upright activity based on physical therapy assessments (e.g., AMPAC-6 clicks or JH-HLM)
5. English or Spanish-speaking
6. Able to provide written informed consent (or via a legally authorized representative if applicable)
7. Meets ORE frame limitations (height = 5'2" to 6'4" and weight ≤ 220 lbs.)

Exclusion Criteria:

1. Cognitive or behavioral impairment that interferes with safe participation [e.g., active delirium (positive CAM-ICU score) or unable to follow commands].
2. Moderate vasopressor or inotrope requirements, including:

   >0.10 mcg/kg/min of norepinephrine >0.03 mcg/kg/min of epinephrine >80.0 mcg/kg/min of phenylephrine >0.04 units/min of vasopressin >5.0 mcg/kg/min of dobutamine >5.0 mcg/kg/min dopamine >0.50 mcg/kg/min of milrinone Any combination of > 3 of any of these, regardless of dose, unless deemed acceptable at the discretion of the treating attending.
3. Sustained ventricular arrhythmias that require intervention at the time of upright mobilization.
4. Any active dose of angiotensin II
5. Positive end-expiratory pressure (PEEP) ≥ 10 cm H20).
6. Except for those with a femoral arterial balloon pump, all patients with existing femoral arterial lines at the time of ambulation are ineligible. However, patients with femoral intraortic balloon pump (IABP) may be considered if, in the judgment of the attending physician and physical therapy team, patient is appropriate for ambulation given patient's clinical status and IABP site and securement status, and if ambulation of appropriate patients with femoral IABP is consistent with local standard of care at the time of ambulation.
7. Skin disintegrity in proximity to the ORE frame
8. Participation in another interventional study that may confound outcome measures.
9. Pregnancy
10. Any other condition that, in the judgment of the clinical or research team, would pose an unacceptable risk or interfere with study participation or interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to ambulation | From the date of ICU admission until the date of first documented upright ambulation session, up to 12 months.
  Time from admission in the ICU to the first upright ambulation session (in hours), assessed up to 12 months from admission.
Ambulation dosage | From first ambulation session through study completion, expected to be less than 1 year
  Step count, total "up time" (minutes), and "walk time" (minutes) measured during each early-ambulation session

SECONDARY OUTCOMES:
Adverse events of special interest | From first ambulation session through study completion, expected to be less than 1 year
  Predefined events considered of particular concern to study safety and tolerability, specifically: discontinuation of a therapy session due to acute medical deterioration (e.g., hypotension, arrhythmia, respiratory distress), pain limiting progression, new requirement for escalation of vasopressor/inotropic support during or immediately after ambulation, unanticipated device-related complication directly linked to the Overground Robotic Exoskeleton or ambulation activity.
Feasibility of Overground Robotic Exoskeleton Early Ambulation (ORE-EA) -1 | From first ambulation session through study completion, expected to be less than 1 year
  Number of staff required to deliver early-ambulation sessions (i.e., set-up, intervention delivery, and take-down)
Feasibility of Overground Robotic Exoskeleton Early Ambulation (ORE-EA) -2 | From first ambulation session through study completion, expected to be less than 1 year
  Role(s) of staff required to deliver early-ambulation sessions (i.e., set-up, intervention delivery, and take-down)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Institute for Rehabilitation, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There currently is no plan to share IPD